CLINICAL TRIAL: NCT01377311
Title: Phase 1 Study of Cornea Stem Cells Cultured on Amniotic Membrane Transplanted on Patients Suffering From Corneal Stem Cell Insufficiency
Brief Title: The Application of Cultured Cornea Stem Cells in Patients Suffering From Corneal Stem Cell Insufficiency
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: We didn't use this tech in patient.
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Wei-Li Chen/Assistant Professor, National Taiwan University, Department of Ophthalmology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 32MD02
Record Dates: First submitted 2011-04-21; First posted 2011-06-21 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Unilateral Limbal Stem Cell Insufficiency
Keywords: limbal stem cell; amniotic membrane; ex vivo expansion of autologous limbal stem cell; unilateral limbal stem cell insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Patients suffering from unilateral limbal stem cell insufficiency. Remove the abnormal surface tissue on the lesion cornea, transplant the amniotic membrane with cultured limbal stem cells on the denuded cornea. Cover with contact lens after operation, and apply topical antibiotics and steroids.
  Interventions: Procedure: Transplant of cultured limbal stem cells on cornea

INTERVENTIONS:
Procedure: Transplant of cultured limbal stem cells on cornea — Remove the abnormal surface tissue on the lesion cornea, transplant the amniotic membrane with cultured limbal stem cells on the denuded cornea. Cover with contact lens after operation, and apply topical antibiotics and steroids.

SUMMARY:
Name of the project：The application of cornea stem cells cultured on amniotic membrane in patients suffering from corneal stem cell insufficiency

Purpose: To develop the technique of using ex vivo expansion of autologous limbal stem cell cultured on amniotic membrane for treatment of patients suffering from limbal stem cell insufficiency

DETAILED DESCRIPTION:
Materials and Methods:

1. Patients suffering from unilateral limbal stem cell insufficiency will be chosen. Make sure those volunteers understand the benefits and risk factors of the operation.
2. Prepare human amniotic membrane, and culture the membrane at37°C，5% CO2，95% room air.
3. One month before transplantation, take 1-2mm2 of limbal tissues from the healthy eye, and culture the limbal tissue on amniotic membrane with 1.5 ml supplemental hormonal epithelial medium (in 5%的 fetal calf serum)
4. Keep culturing the cells in Dulbecco's modified Eagle's medium/Ham's F12 (1:1 ratio), added with 5 % dimethyl sulfoxide, 2 mg/ml human epidermal growth factor ,5 ug/ml insulin, 0.5 ug/ml hydrocortisone, 50 ug/ml gentamicin, 1.25 ug/ml amphotericin B, 5% autoserum。Two to three weeks later, transplantation will be performed after the cells reaches 2-3 cm2
5. Remove the abnormal surface tissue on the lesion cornea, transplant the amniotic membrane with cultured limbal stem cells on the denuded cornea. Cover with contact lens after operation, and apply topical antibiotics and steroids.
6. Postoperatively, observe the patients for one week. After discharge, follow up the patients one week, two week, one month, two months, three months, six months and one year later.
7. Pictures will be taken and the extent of corneal epithelium regeneration, visual acuity, and complications will be recorded during follow-up visits.
8. The investigators plan to collect 20 patients from 1 July,2007 to 30, June, 2010

ELIGIBILITY:
Inclusion Criteria:

* unilateral limbus defect larger than 180 degrees
* repeated corneal epithelial ulcer, loss of visual acuity or neovascularization due to limbal stem cell insufficiency
* no improvement after medical intervention for more than 6 months
* the patient is willing to receive surgery and postoperative follow up

Exclusion Criteria:

* bilateral limbus defect
* limbal stem cell insufficiency does not induce repeated corneal epithelial ulcer, loss of visual acuity or neovascularization
* corneal neovascularization deeper than 1/2 depth of surface matrix
* peripheral surface matrix is less than 200um thick
* no corneal reflex was induced by fiber less than 5mm length measured by Cocet-Bonnet esthesiometer
* improvement under medication
* perisurgical follow up less than 6 months
* unable to be long term followed up postoperatively
* glaucoma patients underwent glaucoma surgery, under medication, IOP > 21mmHg
* glaucoma patients underwent glaucoma surgery, under medication, IOP < 21mmHg, optic disc depression > 90%
* severe incomplete eyelid closure
* severe dye eye syndrome, Schirmer test 5 min < 3 mm
* contralateral eye limbus tissue cannot be obtained, or unable to be cultured
* pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The extent of corneal epithelium regeneration | one week, two week, one month, two months, three months, six months and one year later

SECONDARY OUTCOMES:
visual acuity | one week, two week, one month, two months, three months, six months and one year later
complications | one week, two week, one month, two months, three months, six months and one year later

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Chen, MD, PhD, Principal Investigator — National Taiwan University Hospital, department of Ophthalmology
Locations (1):
- National Taiwan University Hospital, department of Ophthalmology, Taipei, Taiwan